CLINICAL TRIAL: NCT06211244
Title: Association of Serum Eotaxin Levels and Markers of Myocardiac Injury in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Tungs' Taichung Metroharbour Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 112062
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Myocardium; Injury; Coronary Artery Disease
Keywords: coronary artery disease; Eotaxin-1; hemodialysis patients; myocardial injury
MeSH Terms: conditions — Wounds and Injuries; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

Cardiovascular disease (CVD) is one of the leading causes of morbidity and mortality among dialysis patients. Eotaxin-1(also known as Eotaxin and CCL11), an eosinophil-specific chemoattractant that plays a role in a variety of pathologic conditions including allergy, coronary heart disease, and inflammatory bowel disease. CCL11 has been shown to be overexpressed in human atherosclerotic lesions. Moreover, eotaxin-1 levels are higher in non-uremic coronary artery disease patients than in healthy individuals.

Methods:

The study will enrolled 400 hemodialysis patients. Patients are diagnosed with coronary artery disease based on clinical presentation and confirmed by angiography. Serum eotaxin-1 and 8-isoprostane levels are determined by enzyme-linked immunosorbent assay (ELISA). High-sensitivity cTnI immunoassays and albumin redox state by high-performance liquid chromatography are used for measurements.

Aim:

In this study, we aimed to determine the eotaxin-1 concentrations of patients with coronary artery disease and to investigate the role of eotaxin-1 and markers of myocardial injury.

DETAILED DESCRIPTION:
Study Design and Patient Population This cross-sectional trial, and will be carried out in accordance with the Declaration of Helsinki and applicable regulations. The protocol will be sent to the institutional ethics committee and patients' written informed consent will be obtained. To be included in the study, patients will be at least 20-years-old and on outpatient HD for at least 3 months. All the patients were dialyzed three times a week with a high-flux membrane and bicarbonate dialysate solutions. Patients will excluded if they had an acute infection or malignancy. A total of 400 long-term HD patients are randomly invited and enrolled in the study. The medical records will thoroughly reviewed for each subject by a collaborating physician in the study. Information such as underlying kidney disease, cardiovascular disease history, and other comorbid illnesses are abstracted. A pre-existing history of CVD was defined as a history of CAD ( including a history of myocardial infarction, coronary artery angioplasty/stenting/bypass surgery, carotid endarterectomy/stenting), cerebrovascular disease (CVD, e.g., stroke), non-traumatic lower extremity amputation, and lower limb artery bypass surgery/angioplasty/stenting

Measurements Predialysis blood samples are obtained on a mid-week day.Within 30 min after sampling, the remaining blood arecentrifuged at 3,000 g for 10 min, immediately aliquoted and frozen at-80 °C until further analysis. The total serum cholesterol is measured through the reaction of cholesterol esterase/cholesterol oxidase/peroxidase, using Hitachi 747 (Hitachi, Bohemia, NY, USA). HDL cholesterol is quantified after precipitation with polyethylene glycol at room temperature. Serum glucose concentrations are measured by the glucose oxidase method. Low-density lipoprotein cholesterol was calculated using the Friedewald formula. Total serum triglycerides were measured through the reaction of glycerol/ phosphate/oxidase and peroxidase. The serum levels of high-sensitivity C-reactive protein (hsCRP) are measured using a Behring Nephelometer II (Dade Behring, Tokyo, Japan). Serum levels of IL-6 and MCP-1 are measured by a commercially available enzyme-linked immunosorbent assay (Quantikine HS Immunoassaykit, R&D System, Minneapolis, MN, USA). Serum 8-isoprostane concentrations were measured using the ELISA assay (Cayman Chemical, Ann Arbor, Michigan, USA) with a detection limit of 3 pg/mL, according to the manufacturer's instruction.

Serum eotaxin levels will be determined using a commercial ELISA kit (R&D systems, Minneapolis, MN, USA)according to the manufacturer's protocol. In brief, mouse antihuman antibody against eotaxin is used to capture eotaxin from plasma. Captured eotaxin is detected with biotynilated goat antihuman eotaxin antibody. After washing, plates are incubated with streptavidin-HRP, developed with appropriate substrate, and OD450 is determined using an ELISA plate reader. Measurements are done in duplicate in an assay able to detect 10 pg of eotaxin/ml. The intraand inter-assay coefficients of variation values are <4% and <6%, respectively.

The Siemens Atellica IM High Sensitivity Troponin I assay (Siemens Healthineers) is a three-site sandwich immunoassay with a limit of detection of 1.6 ng/L and limit of quantification of 2.5 ng/L. The upper reference limit 99th centile was determined in 2007 samples from healthy individuals as 34 ng/L in women, and 53 ng/L in men, with a single threshold of 45 ng/L. In the reference range population, 75% of patients had values greater than the limit of detection. All measurements were undertaken at a central laboratory, who were blinded to all clinical information with results provided to the research team and linked to the trial database for analysis.

The redox state of serum albumin was determined by fractionating it into human mercaptalbumin (HMA), human nonmercaptalbumin-1 (HNA-1), and human non-mercaptalbumin-2 (HNA-2) with high-performance liquid chromatography (HPLC).

ELIGIBILITY:
Inclusion Criteria:

1. Both sexes aged 20 years or over
2. Received stable hemodialysis at least 3 months.
3. Written informed consent.

Exclusion Criteria:

* acute infection or malignancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients have to be at least 20-years-old and on outpatient hemodialysis (HD) for at least 3 months.
Sampling Method: Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Analysis of biomarkers of serum eotaxin levels. | 1 years
  Eotaxin levels and the serum levels of markers of myocardial injury as well as oxidative stress in a group of prevalent hemodialysis patients.

SECONDARY OUTCOMES:
Redox state of serum albumin assays | 1 years
  The redox state of albumin was determined from serum samples with high-performance liquid chromatography
Analysis of biomarkers of MCP-1 | 1 years
  The MCP-1 was determined from serum samples using standardized enzymelinked immunosorbent assay (ELISA) methods
Analysis of biomarkers of IL-6 | 1 years
  The IL-6 was determined from serum samples using standardized enzymelinked immunosorbent assay (ELISA) methods
Analysis of biomarkers of 8-isoprostane | 1 years
  The 8-isoprostane was determined from serum samples using standardized enzymelinked immunosorbent assay (ELISA) methods
Analysis of biomarkers of High Sensitivity Troponin I | 1 years
  The Siemens Atellica IM High Sensitivity Troponin I assay (Siemens Healthineers) is a three-site sandwich immunoassay with a limit of detection of 1.6 ng/L and limit of quantification of 2.5 ng/L.

CONTACTS AND LOCATIONS:
Overall Officials: Paik Seong Lim, PhD, Principal Investigator — Tungs' Taichung Metroharbour Hospital
Locations (1):
- Tungs' Taichung MetroHarbour Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No